CLINICAL TRIAL: NCT00527267
Title: A Phase 3 Study to Assess the Efficacy and Safety of an Oral Calcimimetic Agent (AMG 073) in Secondary Hyperparathyroidism of End Stage Renal Disease Treated With Hemodialysis
Brief Title: Safety and Efficacy Study of AMG 073 in Hemodialysis Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20000183
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2009-01-26 (Estimated); Status verified 2009-01

CONDITIONS: Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AMG 073 (Experimental): AMG 073
  Interventions: Drug: AMG 073
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 30 mg placebo once daily orally 60 mg placebo once daily orally 90 mg placebo once daily orally 120 mg placebo once daily orally 180 mg placebo once daily orally
  Arms: Placebo
Drug: AMG 073 — 30 mg AMG 073 once daily 60 mg AMG 073 once daily 90 mg AMG 073 once daily 120 mg AMG 073 once daily 180 mg AMG 073 once daily
  Arms: AMG 073

SUMMARY:
Subjects on Hemodialysis will be randomized to AMG 073 or placebo. The screening period is a maximum of 30 days followed by a 26-week treatment period. Lab assessments will be completed throughout the study along with PRO assessments.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women greater than or equal to 18 years of age
* Using effective contraceptive measures
* Mean iPTH during screening of greater than or equal to 300 pg/mL
* Mean calcium during screening of greater than or equal to 8.4 mg/dL
* Stable on hemodialysis

Exclusion Criteria:

* Unstable medical conditions
* Parathyroidectomy within 3 months
* Change in Vitamin D therapy
* Receiving antidepressants
* Experienced an MI within 3 months
* Inability to swallow tablets
* Previously received AMG 073

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2002-02; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of AMG 073 compared with placebo by determining the proportion of subjects with a mean intact parathyroid hormone (iPTH) value <= 250 pg/mL (26.5 pmol/L) during the efficacy assessment phase. | Efficacy Assessment Phase - last 14 weeks of study

SECONDARY OUTCOMES:
To evaluate the efficacy of AMG 073 compared with placebo by determining: the proportion of subjects with a reduction from baseline in iPTH of >= during the efficacy assessment phase | Efficacy Assessment Phase - last 14 weeks of study
To evaluate the efficacy of AMG 073 compared with placebo by determining: percentage change from baseline in calcium x phosphorus (Ca x P) during the efficacy assessment phase | Efficacy Assessment Phase - last 14 weeks of study
To evaluate the efficacy of AMG 073 compared with placebo by determining: changes in self-reported cognitive function from baseline to the end of the efficacy assessment phase | Efficacy Assessment Phase - last 14 weeks of study
To evaluate the safety of AMG 073 compared with placebo. | Entire study - 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_38_AMG_073_20000183.pdf
- See also: FDA-approved Drug Labeling — http://www.sensipar.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com